CLINICAL TRIAL: NCT02238080
Title: Inflammatory Markers and Mircera® Prospective Assessment of Correlation (IMPACT): A Multi-Center Observational Study Investigating the Correlation Between Inflammatory Marker Levels and ESA Dosage in CKD Patients on Dialysis Treated With Mircera®
Brief Title: An Observational Study of Methoxy Polyethylene Glycol-Epoetin Beta (Mircera) in Chronic Kidney Disease Participants on Dialysis
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22556
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants with anemia and CKD who are on dialysis therapy, and who initiate erythropoiesis-stimulating agent (ESA) treatment with methoxy polyethylene glycol-epoetin beta or who are on stable methoxy polyethylene glycol-epoetin beta maintenance therapy, will be treated according to the usual standard of care and current best practice guidelines, and will be observed during the study period.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-Epoetin Beta — Methoxy polyethylene glycol-epoetin beta will be administered according to the usual standard of care and current best practice guidelines and will be observed during the study period.
  Other Names: Mircera®

SUMMARY:
This observational, multi-center, open-label, prospective study will evaluate the relationship between serum interleukin-6 (IL-6) and C-reactive protein (CRP) levels and methoxy polyethylene glycol-epoetin beta dosage in participants with chronic kidney disease (CKD) on dialysis. Participants will be recruited who are on stable methoxy polyethylene glycol-epoetin beta maintenance therapy or will initiate therapy with methoxy polyethylene glycol-epoetin beta.

ELIGIBILITY:
Inclusion Criteria:

* CKD participants undergoing dialysis
* Participants initiating ESA treatment with methoxy polyethylene glycol-epoetin beta or participants on stable methoxy polyethylene glycol-epoetin beta maintenance therapy
* Adequate iron status defined as: serum ferritin above or equal to 100 micrograms per liter (mcg/L) or transferrin saturation above or equal to 20 percent (%)

Exclusion Criteria:

* Conditions known to cause inadequate response to ESA treatment
* Anemia other than symptomatic anemia associated with CKD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with CKD on dialysis therapy, either initiating ESA treatment with methoxy polyethylene glycol-epoetin beta or on stable methoxy polyethylene glycol-epoetin beta maintenance therapy. The study is to be conducted in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Israel (18):
  - Haemek Hospital; Nephrology, Afula
  - Barzilai Medical Centre ; Nephrology and Hypertension, Ashkelon
  - Soroka Medical Center; Nephrology, Beersheba
  - Bnai Zion MC; Nephrology, Haifa
  - Carmel Medical Center; Nephrology, Haifa
  - Wolfson MC; Nephrology, Holon
  - Shaare Zedek Medical Center; Nrphrology Dept., Jerusalem
  - Hadassah Medical Orgainastion; Nephrology, Jerusalem
  - Meir Medical Center; Nephrology Dept., Kfar Saba
  - Western Galilee Hospital; Nrphrology Dept., Nahariya
  - EMMS Nazareth; Nephrology, Nazareth
  - Holy Family Hospital; Nephrology, Nazareth
  - Beilinson Medical Center; Nephrology, Petah Tikva
  - Sheba MC; Nephrology, Ramat Gan
  - Rebecca Sief Hospital; Nephrology, Safed
  - Sourasky MC; Dept. of Nephrology, Tel Aviv
  - Poria Hospital; Nephrology, Tiberias
  - Assaf-Harofeh MC; Nephrology, Zrifin

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants with anemia and chronic kidney disease (CKD) who were on dialysis therapy, and who initiated erythropoiesis-stimulating agent (ESA) treatment with methoxy polyethylene glycol-epoetin beta (Mircera) or who were on stable methoxy polyethylene glycol-epoetin beta maintenance therapy, were treated according to the usual standard of care and current best practice guidelines.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Started | 197
Completed | 172
Not Completed | 25
Not completed — Death | 13
Not completed — Treatment interrupted | 6
Not completed — Withdrawal by Subject | 2
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population included all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta after enrollment in the study.
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants with anemia and CKD who were on dialysis therapy, and who initiated ESA treatment with methoxy polyethylene glycol-epoetin beta or who were on stable methoxy polyethylene glycol-epoetin beta maintenance therapy, were treated according to the usual standard of care and current best practice guidelines.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient (r) Between Serum C-Reactive Protein (CRP) Level and Methoxy Polyethylene Glycol-Epoetin Beta Dose
Description: Regression analysis and Pearson correlation were used to calculate the correlation coefficient (r).
Time Frame: Day 1
Population: ITT population. Participants with stable maintenance treatment were included in this analysis. 'Number of participants analyzed' (N) included participants evaluable for this outcome measure.
Measure: Number; unit: correlation coefficient
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 185
correlation coefficient | 0.1485

2. Primary Outcome: Correlation Coefficient (r) Between Serum Interleukin-6 (IL-6) Level and Methoxy Polyethylene Glycol-Epoetin Beta Dose
Description: Regression analysis and Pearson correlation were used to calculate the correlation coefficient (r).
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 185
correlation coefficient | 0.05557

3. Secondary Outcome: Percentage of Participants With Change in Methoxy Polyethylene Glycol-Epoetin Beta Dose at Month 6
Description: Percentage of participants with change in methoxy polyethylene glycol-epoetin beta dose compared to baseline were reported as per the following categories: (a) No change, (b) Dose increase (1 to greater than [>] 200 micrograms per kilogram [mcg/kg]), and (c) Dose decrease (1 to >200 mcg/kg).
Time Frame: Month 6
Population: ITT population. Participants with stable maintenance treatment were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 189
percentage of participants
  No change | 46.5
  Dose increase | 29.9
  Dose decrease | 23.5

4. Secondary Outcome: Change From Baseline in Methoxy Polyethylene Glycol-Epoetin Beta Dose at Month 6
Time Frame: Baseline, Month 6
Population: ITT population. Participants with stable maintenance treatment were included in this analysis. 'Number of participants analyzed' (N) included participants evaluable for this outcome measure. 'Number analyzed' included participants evaluable for individual categories.
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 186
mcg/kg
  Baseline | 175.2 (109.8)
  Change at Month 6: number analyzed (Participants) | 157
  Change at Month 6 | 13.6 (100.6)

5. Secondary Outcome: Serum CRP Level
Time Frame: Baseline, Month 6
Population: ITT population. Participants with stable maintenance treatment were included in this analysis. 'Number analyzed' included participants evaluable for individual categories.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 189
milligrams per liter (mg/L)
  Baseline: number analyzed (Participants) | 185
  Baseline | 13.7 (18.7)
  Month 6: number analyzed (Participants) | 162
  Month 6 | 16.3 (29.3)

6. Secondary Outcome: Serum IL-6 Level
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 189
picograms per milliliter (pg/mL)
  Baseline: number analyzed (Participants) | 185
  Baseline | 15.8 (13.5)
  Month 6: number analyzed (Participants) | 161
  Month 6 | 16.7 (18.9)

7. Secondary Outcome: Correlation Coefficient (r) Between Serum CRP Level and Methoxy Polyethylene Glycol-Epoetin Beta Dose at Month 6
Description: Regression analysis and Pearson correlation were used to calculate the correlation coefficient (r).
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 155
correlation coefficient | 0.12684

8. Secondary Outcome: Correlation Coefficient (r) Between Serum IL-6 Level and Methoxy Polyethylene Glycol-Epoetin Beta Dose at Month 6
Description: Regression analysis and Pearson correlation were used to calculate the correlation coefficient (r).
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 154
correlation coefficient | 0.19473

9. Secondary Outcome: Predictive Baseline Serum CRP Level for Participants Initiating Treatment With Methoxy Polyethylene Glycol-Epoetin Beta Dose
Time Frame: Day 1
Population: As per change in planned analysis, this outcome was removed due to small sample size and no data was collected for this outcome.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 0

10. Secondary Outcome: Predictive Baseline Serum IL-6 Level for Participants Initiating Treatment With Methoxy Polyethylene Glycol-Epoetin Beta Dose
Time Frame: Day 1
Population: as for outcome 9
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 0

11. Secondary Outcome: Serum Hemoglobin Level
Time Frame: Baseline, Month 6
Population: ITT population. 'Number analyzed' included participants evaluable for individual categories.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 197
grams per deciliter (g/dL)
  Baseline: number analyzed (Participants) | 193
  Baseline | 11.2 (1.0)
  Month 6: number analyzed (Participants) | 171
  Month 6 | 11.2 (1.4)

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months
Description: Safety population included all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta after enrollment in the study.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 48/197
Other Adverse Events (participants affected / at risk) | 15/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=197)
Acute coronary syndrome (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 3
Chills (General disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Localized infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Hemiplegia (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Ischemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Leg amputation (Surgical and medical procedures) | 1
Aortic stenosis (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Microscopic polyangiitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=197)
Anemia (Blood and lymphatic system disorders) | 2
Extrasystoles (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Breast cellulitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Venous pressure increased (Investigations) | 1
Food intolerance (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Leg amputation (Surgical and medical procedures) | 1
Toe amputation (Surgical and medical procedures) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The study was completed as defined in the protocol. Only 197 participants (out of planned 400) were enrolled due to slow recruitment during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.